CLINICAL TRIAL: NCT03846063
Title: Pilot Study Into the Development of an Effective Home-based-exercise-strategy for Patients After THA Delivered on a Tablet-PC
Brief Title: Development of an Effective Home-based-exercise-strategy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Frisius Medisch Centrum (Other); Martini Hospital Groningen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NL50372
Record Dates: First submitted 2019-02-13; First posted 2019-02-19 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Osteoarthritis, Hip; Total Hip Arthroplasty
Keywords: Total hip arthroplasty; Physiotherapy; Osteoarthritis; Usual care; Home-based rehabilitation program
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: A twelve-week home-based exercise strategy will be offered to patients after their discharge from the hospital. This home-based exercise strategy will be delivered by means of videos on a tablet-pc and consist of specified exercise instructions for improving muscle strength, balance and functional movements.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention: Home-based rehabilitation program (Experimental): A twelve-week home-based exercise strategy will be offered to patients after their discharge from the hospital. This home-based exercise strategy will be delivered by means of videos on a tablet-pc and consist of specified exercise instructions for improving muscle strength, balance and functional movements.
  The intervention group will be compared with existing patientdata who received usual care in the Netherlands
  Interventions: Other: Home-based rehabilitation program

INTERVENTIONS:
Other: Home-based rehabilitation program — The duration of the program is 12 weeks. Patients start the program within 7 days after of the surgery. Patients perform exercises independently at home using the tablet PC for instructions. The program includes strengthening and walking exercises based on increasing the muscle force, balance, and functionality. The exercises comprise movements that train abductors, flexors, and extensors of the affected hip. The content of the program is based on previous research and on guidelines from the American Association of Orthopaedic Surgeons. For the rest, the program is designed in line with the most recent guidelines from the Royal Dutch Society for Physical Therapy. Patients are asked to exercise at least 5 days a week, with rest days on Thursday and Sunday. Strengthening exercises will be performed 3 times a week. The instructions for the exercises will be provided by videos on the tablet PC, which patients have to imitate.

SUMMARY:
Osteoarthritis is one of the most common chronic diseases of the musculoskeletal system in elderly. Patients with osteoarthritis experience pain, stiffness and loss of mobility. Due to ageing Western societies in the coming decades the number of elderly with osteoarthritis will progressively increase. Osteoarthritis is a common indicator for a Total Hip Arthroplasty (THA). A hip replacement is one of the most successful orthopedic surgeries. However, with regard to the postoperative rehabilitation a lot can be improved. The current situation after a THA is that physical therapy in the Netherlands is not prescribed by default. Patients are resigned from the hospital and receive home exercises. However, it is not clear whether patients actually carry out these exercises and whether they perform the exercises correctly.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 75 years
* Living independent
* Waiting for THA at either the Martini Hospital Groningen or the Medical Centre Leeuwarden in the Netherlands

Exclusion Criteria:

* Revision surgery
* Medical conditions that disallow independent living
* Cognitive impairment
* Inability to sufficiently read and understand Dutch
* Participating in another rehabilitation program

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Adherence of a home-based rehabilitation program | 12 weeks
  Adherence to the rehabilitation program will be evaluated on the basis of the completion of the planned exercises.
Patient experience of a home-based rehabilitation program at week 4 | 4 weeks
  Patient experience will be done in week 4 (T1) with a questionnaire adapted from the sensing and action to support mobility in ambient assisted living subject evaluation form [12,13]. The questionnaire contains questions about the user experience, the perceived intensity of the intervention, coaching, wearing of the sensor, and acceptability of the technology.
Patient experience of a home-based rehabilitation program at week 12 | 12 weeks
  Patient experience will be done at week 12 at the end of the program (T2) with a questionnaire adapted from the sensing and action to support mobility in ambient assisted living subject evaluation form [12,13]. The questionnaire contains questions about the user experience, the perceived intensity of the intervention, coaching, wearing of the sensor, and acceptability of the technology.

SECONDARY OUTCOMES:
Change in mobility (objective measurement (TUG)) | 6 months
  To assess mobility objectively, the Timed Up & Go test (TUG) will be performed. The TUG is an accepted test to measure mobility. During the TUG, participants will be instructed to stand up from the chair, walk three meters, turn around, walk back and sit down on the chair again. Participants will be asked to walk at a fast but safe pace. The test will be performed three times. The TUG is considered reliable and practical. Measurements will be taken preoperatively (T0) and postoperatively at 4 weeks (T1), 12 weeks (T2) and 6 months (T3).
Change in functional status (objective measurement (FTSST)) | 6 months
  To assess functional status objectively, the Five Times Sit-to Stand Test (FTSST) will be performed. The FTSST is a clinical test to assess lower extremity power and balance. For the FTSST, participants will be asked to stand up and sit down five times at a fast speed. Subjects will be instructed to perform the test with arms crossed in front of the abdomen when possible. The test was performed twice. The FTSST shows good reliability and validity. Measurements will be taken preoperatively (T0) and postoperatively at 4 weeks (T1), 12 weeks (T2) and 6 months (T3).
Change in functional status and hip-related quality of life (self-reported measurement (HOOS)) | 6 months
  The self-reported Hip disability and Osteoarthritis Outcome Score (HOOS) will be used as a disease-specific outcome measure of functional status and quality of life. The HOOS consists of five subscales: pain, other symptoms, function in activities of daily living, function in sport and recreational activities, and hip-related quality of life. Standardized response options are given and each question is scored from 0-4 (on a 5-point Likert scale). A normalized score, ranging from 0-100, will be subsequently calculated for each subscale (0 indicating extreme symptoms and 100 no symptoms). The Dutch version has been proven valid and reliable. Measurements will be taken preoperatively (T0) and postoperatively at 4 weeks (T1), 12 weeks (T2) and 6 months (T3).
Change in health-related quality of life (self-reported measurement (SF-36)) | 6 months
  To measure health-related quality of life, the Short Form 36 (SF-36) will used. The SF-36 is a widely used generic health status questionnaire consisting of 36 questions, divided into eight health concepts: physical functioning, role limitations due to physical problems, social functioning, bodily pain, general mental health, role limitations due to emotional problems, vitality, and general health perceptions. Each raw scale score will be transformed into a linear 0-100 scale. The higher the score, the less disability. In this study only the subscales physical functioning, role limitations due to physical problems, and general health perceptions were analyzed. The SF-36 has proven to be practical, reliable and valid within a general and chronic disease population. Measurements will be taken preoperatively (T0) and postoperatively at 4 weeks (T1), 12 weeks (T2) and 6 months (T3).
Change in health-related quality of life (self-reported measurement (EQ-5D-3L)) | 6 months
  To measure health-related quality of life, the EuroQol 5 Dimensions 3 Level Questionnaire (EQ-5D-3L) will used. The EQ-5D-3L has five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension is divided into three degrees of severity: no problem, some problems and major problems. Actual quality of life will also be identified on the EQ-5D-3L Visual Analogue Scale. Measurements will be taken preoperatively (T0) and postoperatively at 4 weeks (T1), 12 weeks (T2) and 6 months (T3).

CONTACTS AND LOCATIONS:
Overall Officials: Martin Stevens, PhD, Principal Investigator — University Medical Center Groningen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wijnen A, Hoogland J, Munsterman T, Gerritsma CL, Dijkstra B, Zijlstra WP, Dekker JS, Annegarn J, Ibarra F, Slager GE, Zijlstra W, Stevens M. Effectiveness of a Home-Based Rehabilitation Program After Total Hip Arthroplasty Driven by a Tablet App and Remote Coaching: Nonrandomized Controlled Trial Combining a Single-Arm Intervention Cohort With Historical Controls. JMIR Rehabil Assist Technol. 2020 Apr 27;7(1):e14139. doi: 10.2196/14139. PMID 32338621